CLINICAL TRIAL: NCT01611727
Title: Phase II Open-Label, Non-Randomized Trial of Cisplatin Chemotherapy in Patients With BRCA1-Positive Metastatic Breast Cancer
Brief Title: Open-Label,Non-Randomized Trial of Cisplatin Chemotherapy in BRCA1-Positive Metastatic Breast Cancer Patients
Acronym: Cisplatin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pomeranian Medical University Szczecin (Other)
Collaborators: Maria Sklodowska-Curie National Research Institute of Oncology (Other)
Responsible Party: Principal Investigator, Tomasz Byrski, MD, PhD, MD, PhD, Pomeranian Medical University Szczecin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BN-001/83/07
Record Dates: First submitted 2012-05-31; First posted 2012-06-05 (Estimated); Last update posted 2012-07-12 (Estimated); Status verified 2012-07

CONDITIONS: BRCA1 Mutation; Metastatic Breast Cancer
Keywords: BRCA1; survival; metastatic disease; cisplatin
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cisplatin (Experimental)
  Interventions: Drug: Cisplatin

INTERVENTIONS:
Drug: Cisplatin — Cisplatin chemotherapy will be administered as a 75 mg/m2 intravenous (IV) infusion every 3 weeks, for six cycles. Dexamethasone (8mg) will be administered once daily for three days after chemotherapy. Ondansetron (Zofran™) will be used for anti-nausea prophylaxis.

SUMMARY:
Among women with a BRCA1 mutation and breast cancer, choice of chemotherapy is a critical issue. There are emerging data which suggest that mutation carriers may respond differently than non-carriers to particular agents. BRCA1-associated cancers differ from non-hereditary cancers for a range of pathologic and molecular factors, including tumor grade and histologic appearance. Several studies have shown that the response to treatment for women with a BRCA1-associated breast cancer reflects the underlying tumor biology, in particular, the impairment of the DNA damage response and repair pathways, and that it is possible to exploit the sensitivity of BRCA1-associated cancers to DNA damage.

It is equally important that the investigators evaluate the benefit of cisplatin in women with disseminated breast cancer, including those who have previously been treated with one or more chemotherapy regimens. This study is undertaken to evaluate the efficacy of cisplatin chemotherapy in BRCA1 carriers with metastatic breast cancer. The primary objective is to determine the objective response rate of cisplatin in BRCA1 carriers with metastatic breast cancer. The secondary objectives are to determine 3-year survival and to evaluate the toxicities of cisplatin in BRCA1 carriers with metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged ≥ 18 years, with measurable (defined by Response Evaluation Criteria in Solid Tumors (RECIST) criteria (14)) metastatic (stage IV) breast cancer, and who are known to carry a BRCA1 mutation, are eligible.
* In addition, the following are required:

  * adequate hematologic
  * renal, and hepatic function
  * adequate recovery from recent surgery and/or radiation therapy
  * recovery from all prior treatment-related toxicities (to grade < 2 according to National Cancer Institute Common Toxicity Criteria, Version3.0, except alopecia)
  * life expectancy of at least 12 weeks
  * Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1. -
* Patients could have received up to four prior chemotherapies for metastatic disease.

Exclusion Criteria:

* Patients with known brain metastases are not eligible.
* Patients previously treated with a platinum-based chemotherapy are not eligible.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-07; Primary Completion 2009-01 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Tumor Response Rate | Six Months
  This is defined as the percentage of patients who achieved a complete response or partial response by RECIST criteria within the first six months.

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz Byrski, MD, PhD, Principal Investigator — Pomenarian Medical University
Locations (1):
- Pomenarian Medical University, Szczecin, Poland

REFERENCES:
- [Derived] Byrski T, Dent R, Blecharz P, Foszczynska-Kloda M, Gronwald J, Huzarski T, Cybulski C, Marczyk E, Chrzan R, Eisen A, Lubinski J, Narod SA. Results of a phase II open-label, non-randomized trial of cisplatin chemotherapy in patients with BRCA1-positive metastatic breast cancer. Breast Cancer Res. 2012 Jul 20;14(4):R110. doi: 10.1186/bcr3231. PMID 22817698